CLINICAL TRIAL: NCT00297687
Title: A Randomized, Placebo-Controlled, Double Blind, Phase 1 Trial of the Safety, Immunogenicity, and Tolerability of Ascending Doses of Meningococcal Group B rLP2086 Vaccine in Healthy Adults
Brief Title: Study Evaluating the Safety, Immunogenicity and Tolerability of Meningococcal Group B Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 6108A1-500
Record Dates: First submitted 2006-02-24; First posted 2006-02-28 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Meningitis, Meningococcal
Keywords: Vaccines; Healthy Adults; Health; Adult; Meningococcal Vaccines
MeSH Terms: conditions — Meningitis, Meningococcal

INTERVENTIONS:
Biological: MnB rLP2086

SUMMARY:
To determine the safety & immunogenicity of a potential vaccine against meningococcal B disease

ELIGIBILITY:
Inclusion Criteria:

* Healthy 18-25 year olds

Exclusion Criteria:

* Prior history of vaccination with any meningococcal vaccine
* Prior history of any invasive meningococcal disease

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108
Dates: Start 2006-03; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Local & systemic safety throughout the trial

SECONDARY OUTCOMES:
Evidence of an immune response 1 month after dose 2 & 1 month after dose 3

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Australia, medinfo@wyeth.com
Locations (3):
- Australia (3):
  - Herson, Queensland
  - North Adealaide, South Australia
  - Perth, Western Australia